CLINICAL TRIAL: NCT05259475
Title: Ectopic Fat in Singaporean Women - the Culprit Leading to Gestational Diabetes, Metabolic Syndrome, and Type 2 Diabetes
Brief Title: Ectopic Fat in Singaporean Women - the Culprit Leading to Gestational Diabetes, Metabolic Syndrome, and Type 2 Diabetes (TANGO Study)
Acronym: TANGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Collaborators: Wilmar International Limited (Unknown); SATA CommHealth (Singapore) (Unknown); National University Polyclinics, Singapore (Other); National University of Singapore (Other)
Responsible Party: Principal Investigator, Johan Eriksson, Executive Director & Programme Director (Human Development), Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021/00339
Record Dates: First submitted 2022-01-12; First posted 2022-02-28 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both study team and the subjects receiving diet intervention will be blinded on the allocation to food product with or without odd-chain fatty acids (OCFA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle advice alone (Other): The participants in "Lifestyle advice alone" arm (study control) will receive 1 session of diet advice from the study dietitian at the start of the study only. The dietitian will provide dietary advice on the eating plans and instructions for completion of diet checklist. The lifestyle advice on maintaining a healthy diet and regular exercise (~180 mins/ week) will be compatible with recommendations by the Health Promotion Board (Singapore).
  Interventions: Other: Lifestyle Advice
- Diet Intervention (Experimental): Participants will be supplied with 2 main meals per day as part of their daily diet, for 6 days a week. This diet is prescribed as a moderate energy restriction (500-1000 kcal/day) to facilitate weight loss. Additional food products are supplied for breakfast and snacks. Participants will receive individual diet consultations with the study dietitian during the study. Participants are told to consume only low-fat dairy products (milk, yoghurt), and avoid ruminant meat (beef, lamb), cheese, butter, butter-containing food products, and sugar-sweetened beverages.
  Interventions: Other: Diet Intervention
- OCFA Meal-Based Diet-Intervention (Experimental): Participants in the "OCFA meal-based diet-intervention" arm will be provided with OCFA-containing food product, in addition to the lunch and dinner meals (6 days a week) given in the "Diet Intervention" arm. Participants will receive individual diet consultations with the study dietitian during the study. Participants are told to consume only low-fat dairy products (milk, yoghurt), and avoid ruminant meat (beef, lamb), cheese, butter, butter-containing food products, and sugar-sweetened beverages.
  Interventions: Other: OCFA Meal-Based Diet-Intervention

INTERVENTIONS:
Other: Lifestyle Advice — Maintain a weekly healthy diet and regular exercise.
  Arms: Lifestyle advice alone
Other: Diet Intervention — Calorie-restricted meals (lunch and dinner)
  Arms: Diet Intervention
Other: OCFA Meal-Based Diet-Intervention — OCFA-containing food product
  Arms: OCFA Meal-Based Diet-Intervention

SUMMARY:
Ectopic fat is the accumulation of adipose tissue in anatomical sites not classically associated with fat storage - for example, in the liver and skeletal muscles. Excessive fat accumulation in liver cells, often diagnosed as non-alcoholic fatty liver disease (NAFLD), is a precursor to a wide range of liver conditions and metabolic disorders. The usual standard of care for NAFLD is to advise weight loss through controlled diet and physical activity, but the outcome of weight management and treatment of NAFLD is highly variable.

Diet interventions - such as the Mediterranean, ketogenic, paleo, and high-protein-low-carbohydrate diets - have shown varied benefits in the management of NAFLD. However, food-based interventions must align with cultural and regional preferences in food to succeed in making the modifications part of the habitual diet. A recent diet intervention study (Della Pepa et al., 2020) highlighted that the components of a diet, rather than its caloric content, play a greater role in achieving healthier outcomes. In this study, a multifactorial diet intervention using locally sourced and produced meals will be implemented with the aim of reducing elevated liver fat content in healthy women diagnosed with NAFLD.

The study will also evaluate the effects of the proposed diet on the participants' metabolic health and describe potential changes in their gut microbiome signatures (via frequent stool samples). The dysregulation of the gut microbiota has been linked to the development of NAFLD and it is known that the composition of the gut microbiota could be modified by dietary intake. This study will investigate the association of gut microbiome signatures with elevated liver fat in Asian women and test whether the dietary intervention will modify their gut microbiota.

Finally, ectopic fat in the liver is a highly prevalent condition worldwide but the cut-off values for NAFLD has been largely derived from studies performed in Western populations. This study seeks to cross examine the diagnostic ranges in various clinical assessments of NAFLD that commonly involve ultrasound spectroscopy (Fibroscan), fatty liver indexes (FLI) and magnetic resonance spectroscopy (MRS). This effort seeks to derive appropriate cut-off values for NAFLD in Singaporean-Chinese women.

DETAILED DESCRIPTION:
The study will consist of a 12-week, parallel three-arm, single-centre, randomized controlled trial (RCT); 90 women of Chinese ethnicity matched for age and BMI will be randomized to one of 3 study arms in 1:1:1 ratio by Blockrand R software at Week -1 visit. The study arms are: (1) Lifestyle advice alone, (2) Lifestyle advice with calorie-restricted diet-intervention, and (3) Lifestyle advice with calorie-restricted diet-intervention inclusive of odd-chain fatty acids (OCFA)-containing food product.

In all 3 study arms, the lifestyle advice on maintaining a healthy diet and regular exercise (~180 mins/ week) will be compatible with recommendations by Health Promotion Board. The participants in the control study arm (Lifestyle advice alone) will receive 1 session of diet advice from the study dietician at the start of the study only. The dietitian will provide dietary advice on the eating plans and instructions for completion of diet checklist.

In the "Diet Intervention (calorie-restricted multifactorial diet)" study arm (arm 2), a moderate energy restriction (500-1000 kcal/day) will be prescribed to facilitate weight loss. To facilitate compliance, participants in the diet-intervention arms will receive individual diet consultations with the study dietitian during the study. Participants in both the meal-based diet-intervention arms (arm 2 and arm 3) will be supplied with 2 main meals per day as part of their daily diet, for 6 days a week. Additional food products may be supplied for breakfast and snacks. The diet will be designed to be nutritionally replete, feasible, and sustainable in the long-term. The diet will be based on whole grain-based products, vegetables, legumes, extra virgin olive oil, fruits, almonds, salmon, and plant-based meat analogues. Diet plans will be individualized and energy matched to enable any metabolic differences between arms to be attributed to the macronutrient profiles of the diets, without confounding by differences in weight loss between diet arms. Energy requirements will be calculated by indirect calorimetry (Quark CPET, COSMED) with an activity factor.

Participants in the "OCFA meal-based diet-intervention" study arm (arm 3) will be provided with a daily OCFA-containing food product, in addition to the lunch and dinner meals. Both the participants in arm 2 and 3 will be receiving the same lunch and dinner meals. Participants in both the meal-based diet-intervention arms (arm 2 and arm 3) will be told to consume only low-fat dairy products (milk, yoghurt), avoid ruminant meat (beef, lamb), avoid cheese, butter and butter-containing food products. Both diet-intervention arms will be told to avoid sugar-sweetened beverages.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* Females, Age 21-45 years
* Body mass index (BMI) 23-35 kg/m2
* Not planning to conceive within 6 months from enrolment
* Elevated liver fat content (FibroScan CAP score >=268 dB/m)

Exclusion Criteria:

* Do not intend to reside in Singapore for the next 6 months
* Delivered within the last 6 months
* Currently pregnant or breastfeeding
* Having more than 5% weight loss over the past 3 months
* Receiving antibiotics or suffering from diarrhoea over the last 3 months
* Not willing to adhere to lifestyle intervention required by study
* Following special diets or having intentional dietary restrictions (e.g. vegetarians/vegans/ketogenic diet)
* Having contraindications for MRI e.g. metallic implants such as cardiac pacemaker
* Having alcohol consumption on more than 4 days per week with 6 or more alcoholic drinks per week
* Current and/or history of diabetes mellitus, other than GDM (Gestational Diabetes Mellitus)
* Having chronic medical conditions such as cancer, severe gastrointestinal disorders, infectious diseases such as hepatitis and severe mental disorders
* Having uncontrolled hypertension (> 150/90 mmHg)
* Having any medication and/or supplements which may interfere with study results
* Having allergies or intolerances to any common food ingredients including eggs, fish, milk, sesame, mustard, sulphites, peanuts and tree nuts, shellfish, soy, wheat, gluten, cereal, fruits, dairy products, meat, vegetable, sugar and sweetener, food colourings or flavourings, etc.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in liver fat content. | Screening, and Week 12
  Assessed by Fibroscan CAP (Controlled Attenuation Parameter) score.

SECONDARY OUTCOMES:
Change in liver fat, intramyocellular lipid content (IMCL), and abdominal fat compartments. | Week 0, and 12
  MRI/MRS will be used to measure the amount of fat in the liver, abdomen and leg of the participants.
Change in insulin sensitivity and Fatty Liver Indexes (FLI). | Week 0, 4, 8 and 12
  Fatty Liver Indexes (FLI) will be calculated based on blood measurements of liver enzymes, lipids, and insulin.
Change in sleep quality as assessed by the OURA Ring Sleep Score. | Week 0, and 12
  Participants will be issued a wearable device to capture durations of deep sleep, rapid eye movement (REM) sleep, light sleep, and nightly heart rate. Sleep Score ranges from 0-100, where a higher score reflects better sleep outcome.
Change in daily physical activity levels as assessed by the OURA Ring Activity Score. | Week 0, and 12
  Participants will be issued a wearable device to capture durations of activity, inactivity and rest. Activity Score ranges from 0-100, where a higher score reflects better balance between activity and rest.
Change in quality of life. | Week 0, 4, 8 and 12
  Assessed by the 36-Item Short Form Survey (SF-36).
Change in anxiety (if any). | Week 0, 4, 8 and 12
  Assessed by State-Trait Anxiety Inventory (STAI).
Change in depression (if any). | Week 0, 4, 8 and 12
  Assessed by Beck Depression Inventory-II (BDI-II).
Change in the composition of gut microbiota from baseline due to the diet intervention. | Week 0, 2, 4, 8, and 12
  Assessed using gut metagenome and metatranscriptome profiling.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Development Research Centre (Hdrc), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chooi YC, Magkos F, Yaligar J, Michael N, Sadananthan SA, Kway YM, Velan SS, Lim KJ, Lai X, Wong LH, Chong YS, Loo EXL, Eriksson JG. Adherence to a "MediterrAsian" diet is associated with weight loss-independent improvements in liver fat and lipid profile, but not glucoregulation or inflammation: secondary analysis of a randomized controlled trial. Front Nutr. 2025 Jul 24;12:1623612. doi: 10.3389/fnut.2025.1623612. eCollection 2025. PMID 40777170
- [Derived] Salamanca-Sanabria A, Chooi YC, Loo EXL, Lai X, Volchanskaya VSB, Chong YS, Eriksson JG. Potential effects of Asian-adapted Mediterranean diet in depression and anxiety among women with metabolic dysfunction-associated steatotic liver disease: a secondary analysis. Front Nutr. 2025 Jul 8;12:1589412. doi: 10.3389/fnut.2025.1589412. eCollection 2025. PMID 40697557
- [Derived] Chooi YC, Zhang QA, Magkos F, Ng M, Michael N, Wu X, Volchanskaya VSB, Lai X, Wanjaya ER, Elejalde U, Goh CC, Yap CPL, Wong LH, Lim KJ, Velan SS, Yaligar J, Muthiah MD, Chong YS, Loo EXL, Eriksson JG; TANGO Study Group. Effect of an Asian-adapted Mediterranean diet and pentadecanoic acid on fatty liver disease: the TANGO randomized controlled trial. Am J Clin Nutr. 2024 Mar;119(3):788-799. doi: 10.1016/j.ajcnut.2023.11.013. Epub 2023 Nov 29. PMID 38035997